CLINICAL TRIAL: NCT05916261
Title: Clinical Study of Personalized Tumor Vaccines mRNA-0217/S001 and Pabolizumab in Patients With Advanced Pancreatic Cancer
Brief Title: Personalized Tumor Vaccines and Pabolizumab in Patients With Advanced Pancreatic Cancer
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022PCV001
Record Dates: First submitted 2023-05-23; First posted 2023-06-23 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-05

CONDITIONS: Advanced Pancreatic Cancer
Keywords: Personalized neoantigen tumor vaccine

STUDY DESIGN:
Intervention Model Description: The traditional 3+3 design will be used in dose escalation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Personalized neoantigen vaccine or neoantigen tumor vaccine + Pembrolizumab (Experimental): In dose escalation phase, subject will only receive personalized neoantigen tumor vaccine. In dose expansion phase, subject will receive personalized neoantigen tumor vaccine combination with Pembrolizumab .
  Interventions: Biological: Personalized neoantigen tumor vaccine

INTERVENTIONS:
Biological: Personalized neoantigen tumor vaccine — neoantigen tumor vaccine with or without Pembrolizumab In dose escalation phase, subjects will receive neoantigen tumor vaccine only. In dose expansion phase, subjects will receive neoantigen tumor vaccine combination with Pembrolizumab

SUMMARY:
The main objective of this study was to observe and evaluate the safety and tolerability of mRNA-0217/S001 vaccine encoding personalized tumor neoantigens alone/in combination with Pembrolizumab injection for the treatment of Advanced Pancreatic Cancer. The secondary objective was to observe the preliminary efficacy of mRNA-0217/S001 personalized tumor vaccine in the treatment of advanced solid tumors with neoantigen-specific CD4+ and CD8+ T lymphocyte responses, objective tumor response rate (ORR) and disease control rate (DCR), progression-free survival (PFS) and overall survival (OS) caused by mRNA-0217/S001 personalized tumor vaccine.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects voluntarily signed written informed consent files,Able to comply with the study protocol, in the investigator's judgment
2. Subjects must be >/= 18 years of age at time of informed consent, regardless of gender
3. Subjects with locally advanced, recurrent or metastatic solid tumors confirmed by histology or cytology within the past 6 months, who have failed standard treatment or are currently not suitable for standard treatment
4. No copy number variations (CNVs) or loss of heterozygosity (Loss-of heterozygosity, LOH) were found in HLA-related genes and chromosomal regions by gene sequencing
5. Advanced or metastatic lesions confirmed by immunohistochemistry, and cryopreserved tissues/cells, enough for WES and RNAseq sequencing, and predicted by bioinformatics analysis, at least one antigen effectively presented by self-HLA was found , such as KRAS or TP53 mutations and correspondingly presented HLA types
6. Life expectancy ≥ 4 months
7. Have measurable disease per RECIST 1.1 as assessed by the local site investigator/radiology. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions
8. Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale
9. Have adequate organand bone marrow function,No use of granulocyte colony-stimulating factor (G-CSF), granulocyte-macrophage colony-stimulating factor (GM-CSF), red blood cell transfusion and platelet transfusion within 14 days before the examination.
10. Fertile eligible patients (male and female) must agree to use reliable contraceptive methods (hormone or barrier method or abstinence) during the trial and at least 90 days after the last dose. female patients of childbearing age before the first dose A blood pregnancy test within 7 days must be negative.
11. Subjects need to undergo virological examination: those without CMV and EBV, HIV, HBV, HCV, and syphilis infection (only in the baseline period)

Exclusion Criteria:

1. Has had chemotherapy, hormone therapy, traditional Chinese medicine, or biological cancer(for mitomycin and nitrosoureas within 6 weeks from the first dose of the drug in this study)， prior to the first dose of study therapytherapy within 4 weeks ,Or within 5 half-lives of immunotherapy, molecular targeted therapy
2. Subjects have undergone major surgical procedures other than the diagnosis or biopsy of the current tumor within 4 weeks before the first dose of mRNA-0217/S001, or are expected to undergo major surgery during the study period
3. Subjects have received allogeneic hematopoietic stem cell transplantation or organ transplantation in the past, or those who plan to receive organ transplantation during this study
4. Subjects have previously received other tumor vaccines or cell therapy
5. Brain metastases with clinical symptoms, spinal cord compression, cancerous meningitis, or other evidence that the brain and spinal cord metastases have not been controlled, and the researchers judged that they are not suitable for enrollment
6. Other malignant tumors known to be progressing or requiring active treatment in the past 2 years (except for non-melanoma skin cancer, superficial bladder cancer, and carcinoma in situ of the cervix that have been cured by surgical curative treatment)
7. History of interstitial lung disease (ILD), pulmonary fibrosis
8. Have a history of serious cardiovascular and cerebrovascular diseases, including but not limited to a) severe cardiac rhythm or conduction abnormalities, such as ventricular arrhythmia requiring clinical intervention, second-third degree atrioventricular block corrected QTc interval male > 450 milliseconds, female > 470 milliseconds, b) Acute coronary syndrome, congestive heart failure, aortic dissection, stroke or other cardiovascular and cerebrovascular events of grade 3 or above occurred within 6 months before the first administration, c) New York Heart Association (NYHA) ≥ III heart failure or left ventricular ejection fraction (LVEF) < 50%.
9. Other serious and/or uncontrollable diseases, which may affect the subject's participation in this study, include but not limited to a) a history of severe drug allergy, or is known to be allergic to any tumor vaccine and pembrolizumab formulation components or has had severe allergic reactions to other monoclonal antibodies in the past, b) A history of immunodeficiency, including HIV positive or other acquired or congenital immunodeficiency diseases, c) Evidence of severe or uncontrolled liver or kidney disease, d) Uncontrolled high blood pressure, diabetes, etc., e) Patients with active ulcers, gastrointestinal bleeding, f) Serious infection requiring intravenous antibiotics or hospitalization or uncontrolled active infection within 4 weeks before the first dose, g) have an active syphilis infection.
10. Participate in other clinical trials within 4 weeks before the first dose (except for screening failure)
11. Those who are currently receiving systemic steroids (except those who have recently or currently used inhaled steroids)
12. Pregnant and lactating women
13. Imaging (CT or MRI) shows that the tumor invades large blood vessels and has a tendency to hemorrhage
14. Have clinically significant thyroid dysfunction, and the investigator judges that they are not suitable for enrollment
15. Active pneumonia found in chest CT scan during the screening period
16. Uncontrolled pleural effusion, pericardial effusion, or ascites that needs repeated drainage
17. Subjects who have adverse reactions of the previous anti-tumor therapy have not recovered to NCI-CTCAE 5.0 grade evaluation ≤ grade 1 (except for hair loss)
18. HBsAg positive and peripheral blood HBV DNA detection value is higher than the upper limit of normal, and/or HCV Ab positive and HCV RNA detection value is higher than the upper limit of normal
19. Researchers believe that there are other reasons that are not suitable for participating in clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-04-26 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) or Dose-limiting toxicity(DLT),If MTD is not reached, Biologically Effective Dose (BED) | Up to 27 weeks
  The highest dose of a drug or treatment that does not cause unacceptable side effects.
Reaction of antigen-specific T cells in peripheral blood | Up to 27 weeks
  mRNA-0217/S001 personalized tumor vaccine induced neoantigen-specific CD4+ and CD8+ T lymphocyte responses
Objective response rate (ORR) | Up to 105 weeks
  ORR calculates the ratio of the number of patients whose best response is complete remission (CR) or partial remission (PR) to the total number of evaluable patients according to RECIST 1.1 criteria. Those who have not been evaluated for lesion and tumor response will be regarded as non-evaluable patients and will not be counted.
Disease control rate (DCR) | Up to 105 weeks
  DCR calculates the ratio of the number of patients whose best response is complete remission (CR), or partial remission (PR), or stable disease (SD) to the total number of evaluable patients according to RECIST 1.1 criteria. Those who have not been evaluated for lesion and tumor response will be regarded as non-evaluable patients and will not be counted.

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | Up to 105 weeks
  During the trial conduction, all adverse events (including laboratory abnormality and clinical events) will be closely monitored, and all ≥ grade 3 adverse events per CTCAE (v 5.0) will be recorded, including but not limited to the toxicities potentially suspected to relate to injection procedures and/or mRNA Tumor Vaccine therapy as listed below:
  Local erythema at the injection site, local allergic reactions at the injection site, fatigue, fever, chills, flu-like manifestations, vomiting, centrocytopenia, other unexpected adverse events
Progression-free survival (PFS) | Up to 105 weeks
  Progression-free Survival of Personalized mRNA Tumor Vaccine
overall survival (OS) | Up to 3 years
  Overall Survival of Personalized mRNA Tumor Vaccine

CONTACTS AND LOCATIONS:
Overall Officials: Baiyong Shen, M.D.&Ph.D, Study Director — Ruijin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine
Locations (1):
- Ruijin-Hainan Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Qionghai, Hainan, China

IPD SHARING:
Plan to Share IPD: No